CLINICAL TRIAL: NCT03291704
Title: PILOT STUDY: The Effect of Thermal Therapy Using a Rechargeable, Wireless Device on Meibomian Gland Dysfunction
Brief Title: Investigating the Effect of At Home Thermal Therapy on Dry Eye Patients With Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMay Care Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Meibomian Gland Dysfunction
Record Dates: First submitted 2017-09-12; First posted 2017-09-25 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Disease
Keywords: Dry Eye; Thermal Therapy; Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thermal Therapy (Experimental): Heat application using at home thermal therapy device
  Interventions: Device: Thermal therapy device

INTERVENTIONS:
Device: Thermal therapy device — Thermal therapy of blocked Meibomian glands
  Other Names: umayREST

SUMMARY:
The purpose of this pilot study is to determine the feasibility of at home thermal therapy with a wireless, portable device, as an effective management of Meibomian Gland Dysfunction.

This will be done by assessing patients for improvement in symptoms and ocular oil gland function after 4 weeks of a daily thermal therapy application.

DETAILED DESCRIPTION:
This study will be a non-randomized, open label study of subjects with documented MGD. All subjects will be sent home with a wireless, portable thermal therapy device and examined pre and post treatment period. Subjects will be asked to use the device at bedtime for 5 minutes daily for 4 weeks. After treatment subjects will be re-examined and measured for clinical and symptomatic change in their MGD as well as changes to their sleep quality and anxiety index. Subjects will also be followed after treatment has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MGD
* Minimum age 18 years

Exclusion Criteria:

* History of ocular disease, trauma, surgery (other than refractive), orbital cancer
* 3 month history of ocular infection and/or ocular inflammation not associated with dry eye
* 3 month history of any active physician administered or prescription dry eye treatment
* Pregnant, potentially pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in Non-Invasive Tear Film Break Up Time (NITFBUT) in Seconds | Before and after 4 weeks of daily treatment
  Ocular surface analysis of tear film evaporation

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Score | Before and after 4 weeks of daily treatment
  Standardized symptom questionnaire
Meibum Expressibility | Before and after 4 weeks of daily treatment
  Grade of Meibum oil expressibility from Meibomian Gland
Sleep Quality | Before and after 4 weeks of daily treatment
  Pittsburg Sleep Quality Index (PSQI)
State Trait and Anxiety | Before and after 4 weeks of daily treatment
  State-Trait Anxiety Index (STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Hermina Strungaru, MD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: Undecided